CLINICAL TRIAL: NCT02991885
Title: A Randomized, Double-blind, Placebo-controlled, Multi-centre Study to Assess the Safety, Tolerability and Immunologic Effects of HAL-MPE1 Subcutaneous Immunotherapy in Adult and Paediatric Subjects With Peanut Allergy
Brief Title: HAL-MPE1 Safety and Tolerability Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: HAL Allergy (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HAL-MPE1/0049
Record Dates: First submitted 2016-11-21; First posted 2016-12-14 (Estimated); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: Peanut Allergy
MeSH Terms: conditions — Peanut Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HAL-MPE1 (Experimental): HAL-MPE1 is an off-white to white liquid suspension containing modified peanut extract
  Interventions: Biological: HAL-MPE1
- HAL-MPE1 placebo (Placebo Comparator): HAL-MPE1 placebo without modified peanut extract
  Interventions: Drug: HAL-MPE1 placebo

INTERVENTIONS:
Biological: HAL-MPE1 — Weekly subcutaneous administrations of HAL-MPE1
  Other Names: Modified peanut extract
  Arms: HAL-MPE1
Drug: HAL-MPE1 placebo — Weekly subcutaneous administrations of HAL-MPE1 placebo
  Other Names: Placebo for modified peanut extract
  Arms: HAL-MPE1 placebo

SUMMARY:
The aim of this study is to confirm safety and tolerability of incremental doses of HAL-MPE1 subcutaneous immunotherapy (SCIT) in peanut allergic adults, and subsequently assess the safety and tolerability in adolescents and children with peanut allergy.

DETAILED DESCRIPTION:
At the time of the study there was no effective treatment available for peanut allergy other than avoidance of peanut allergens. There was high unmet medical need for a disease modifying treatment for peanut allergy, especially for peanut allergic children, since this age group is at highest risk of peanut-related anaphylaxis requiring hospitalization. A chemically modified, aluminum hydroxide adsorbed peanut extract (HAL-MPE1) for subcutaneous administration has been developed. The safety and tolerability of HAL-MPE1 have been established in a First-in-human (FIH) study in adults.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent/assent
* Male or female subjects aged 5- 50 years
* A well-documented medical history of systemic reactions after ingestion of peanut
* Positive serum specific anti-peanut (>5.0 kU/L) and Ara h 2 Immunoglobulin E (IgE)-test (>2.0 kU/L)
* Skin prick test (SPT) to peanut ≥3 mm compared to negative control within the last 2 years
* Forced expiratory volume at first second (FEV1)>80% predicted (adults and adolescents) or Peak expiratory flow(PEF)>80% predicted (children)
* Negative pregnancy test at screening for females of childbearing potential

Females of childbearing age must be using an effective method of contraception to prevent pregnancy and agree to continue to practice an acceptable method of contraception for the duration of participation in the study. Contraceptive measures considered adequate are:

* hormonal contraceptives such as contraceptive pills, transdermal patches, intrauterine device (IUD), intrauterine system (IUS) implant, or vaginal ring (started - least 4 weeks prior to Investigational Medicinal Product (IMP) administration)
* double barrier methods: e.g. condom or occlusive cap (diaphragm or cervical/vault caps) plus spermicidal agent
* surgical sterilization of the female participant (removal of the uterus or ovaries or tubal ligation)
* participants who are postmenopausal (12 consecutive months without a period) for at least 2 years
* male partner sterilization (vasectomy with documentation of azoospermia) prior to the female patient's entry into trial and is the sole sexual partner for that female patient
* sexual abstinence or having no sexual relationship with a man.

Exclusion Criteria:

* Subjects with a history of severe anaphylaxis to peanut with the following symptoms: hypotension, neurological compromise (collapse, loss of consciousness or incontinence) after ingestion of peanuts
* Baseline serum tryptase level >20 µg/l
* Known allergy or hypersensitivity to an excipient in the study drug or placebo
* Clinical features of moderate or severe persistent asthma (as guided by the 2007 NHLBI Guidelines and according to the opinion of the investigator)
* Asthma with FEV1<80% predicted (adults, adolescents) or PEF <80% predicted (children)
* Asthma Control Test (ACT) ≤ 19
* Asthma attack/exacerbation within the last 3 months
* Hospitalization due to asthma within the last year
* Two or more courses of oral steroids within the last 6 months
* History of intubation /mechanical ventilation due to allergies or asthma
* Participation in any interventional study with peanut immunotherapy in the last year
* Any specific immunotherapy (SCIT, Sublingual Immunotherapy (SLIT) or OIT) during the study period
* Severe immune disorders (including autoimmune diseases) and/or diseases requiring immunosuppressive drugs
* Presence of chronic urticaria, atopic dermatitis with flare or atopic dermatitis with SCORAD>40
* Active malignancies or any malignant disease within the past 5 years
* Severe (uncontrolled) diseases that could increase the risk for subjects participating in the study, including but not limited to: any severe or unstable lung diseases; endocrine diseases; clinically significant renal or hepatic diseases, renal impairment, haematological disorders; severe ongoing symptomatic allergic diseases
* History of cardiovascular disease, uncontrolled hypertension or arrhythmias
* Diseases with a contraindication for the use of epinephrine (e.g. hyperthyroidism, glaucoma)
* Use of systemic steroids within 4 weeks before start of the study and during the study
* Treatment with beta-blockers or angiotensin-converting enzyme (ACE) inhibitors
* Vaccination within one week before start of therapy or during study unless considered necessary based on the opinion of the investigator.
* Anti-IgE/anti-Tumor Necrosis Factor (TNF)/omalizumab therapy or any biologic immunomodulatory therapy within the 6 months prior to inclusion and during the study
* Participation in a clinical study with a new investigational drug within the last 3 months or for a biological within the last 6 months prior to or during the study
* For female adolescents and adults of childbearing potential: Pregnancy (test performed at screening), lactation or inadequate contraceptive measures for women of child-bearing age (contraceptive measures considered adequate are: intrauterine devices, hormonal contraceptives, such as contraceptive pills, implants, transdermal patches, hormonal vaginal devices or injections with prolonged release, sexual abstinence or having no sexual relationship with a man)
* Alcohol, drug or medication abuse within the past year
* Any clinically significant abnormal laboratory parameter at screening
* Lack or expected lack of cooperation or compliance
* Unable to use the epinephrine pen correctly
* Severe psychiatric, psychological, or neurological disorders
* Subjects who are employees of the sponsor, institution or 1st degree relatives or partners of the investigators

Ages: 5 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 42 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
Occurrence of local and systemic reactions | within 30 minutes to >4 hours
  Occurrence of immediate (≤ hour), early (1-4) and late (> 4 hours) local and systemic reactions reactions
Occurrence of treatment emergent adverse events | Throughout study completion, an average 16 weeks
  Treatment emergent adverse events will be collected by reporting of adverse events and by clinical relevant changes in laboratory values, vital signs, lung function and aluminum levels in plasma and urine

SECONDARY OUTCOMES:
Changes immunoglobulin levels | Before and after 4, 8 and 16 weeks of treatment
  Serum specific and component specific immunoglobulin levels
Changes in basophil activation | Before and after 16 weeks treatment
  In vitro determination of basophil activation upon antigen stimulation
Changes in histamine release test | Before and after 16 weeks treatment
  Determination of histamine release and total cellular histamine content induced by peanut

CONTACTS AND LOCATIONS:
Overall Officials: Robert Wood, MD, Principal Investigator — John Hopkins Hospital Unversity-Divison of Pediatric Allergy; Scott Sicherer, MD, Principal Investigator — Jaffe Food Allergy Institute, Icahn School of Medicine at Mount Sinai; Edwin Kim, MD, Principal Investigator — UNC Rheumatolory Allergy & Immunology Clinic
Locations (7):
- United States (6):
  - John Hopkins Hospital University-Divison of Pediatric Allergy, Baltimore, Maryland
  - Jaffe Food Allergy Institute, Icahn School of Medicine at Mount Sinai, New York, New York
  - UNC Rheumatolory Allergy & Immunology Clinic, Chapel Hill, North Carolina
  - Allergy, Asthma and Immunology Center, Tulsa, Oklahoma
  - South Texas Allergy & Asthma Medical Professionals (STAAMP), San Antonio, Texas
  - Asthma, Inc., Seattle, Washington
- Inflamax Research Limited, Mississauga, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Reyes AJ, Hosein AS, Ramcharan K, Perot S. Anaphylaxis and other allergic reactions to food: a global challenge. BMJ Case Rep. 2020 May 14;13(5):e231425. doi: 10.1136/bcr-2019-231425. PMID 32414772